CLINICAL TRIAL: NCT05774782
Title: A Prospective, Multi-center, Single Arm Clinical Study to Evaluate the Safety and Effectiveness of the Flow Diverter Stent System in the Treatment of Cerebral Aneurysms
Brief Title: Parent Artery Reconstruction for Cerebral Aneurysms Using a Novel Flow Diverter With Surface Modification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinomed Neurovita Technology Inc. (Industry)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNSC-CFD-202204
Record Dates: First submitted 2023-03-06; First posted 2023-03-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Aneurysm; Cerebral Aneurysm Unruptured
Keywords: flow diverter; endovascular therapy
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cerebral flow diverter (Experimental): The cerebral flow diverter in the endovascular treatment of wide-necked cerebral aneurysms
  Interventions: Device: Cerebral flow diverter

INTERVENTIONS:
Device: Cerebral flow diverter — The surface-modified flow diverter is an intracranial implant designed to be placed in a parent artery so as to divert blood flow away from an aneurysm.

SUMMARY:
The primary objective of this trial is to evaluate the safety and efficacy of the cerebral flow diverter in the endovascular treatment of wide-necked cerebral aneurysms

DETAILED DESCRIPTION:
The investigation is a prospective, multi-center, single arm clinical study. The trial is anticipated to last from March 2023 to January 2025 with 143 subjects recruited in around 10 China centers. The population for this study is subjects with wide-necked intracranial aneurysms who are suitable candidates for flow diverter implantation. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be enrolled after offering informed consent form. The study consists of six visits including preoperative screening, operation date, 7days or at discharge, 30 days, 180 days, and 1 year. The primary efficacy endpoint was complete aneurysm occlusion with parent artery stenosis ≤ 50% at one year post-procedure in the absence of additional treatments, while the primary safety endpoint was no major stroke in the treated artery territory or neurological death at one year post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years to 75 years, male or non-pregnant female.
2. Unruptured wide-necked cerebral aneurysms confirmed by preoperative imaging (Wide-necked is defined as width ≥ 4 mm or a dome-to-neck ratio < 2).
3. Parent vessel with a diameter range of 1.75-6.0 mm.
4. Those who voluntarily participate in the study and sign informed consent form.

Exclusion Criteria:

1. Subject with target aneurysms are blood blister-like aneurysms, pseudoaneurysms, arteriovenous malformation, moyamoya disease-related aneurysm, or multiple aneurysms that cannot be treated with a single stent.
2. Severe arteriosclerosis or tortuosity of intracranial artery, and the device is difficult to reach the target vessel.
3. Subject with target aneurysm previously treated with craniotomy or other endovascular interventional therapy.
4. Known sensitivity to antiplatelet medications, anticoagulant medications, radiographic contrast agents, anesthetic, nickel, platinum-tungsten alloy, platinum-iridium alloy, and poly-N-[Tris(hydroxymethyl)methyl] acrylamide (poly-NTMA).
5. Severe respiratory system, liver and kidney diseases (such as creatinine ≥ 3.0 mg/dL (except dialysis)) or blood coagulation disorders before operation.
6. Platelet count is less than 100×109/L, international normalized ratio (INR) is more than 1.5.
7. Hospitalized surgical treatment within the previous 30 days or planned within the next 180 days after operation.
8. Severe neurological deficit that renders the patient incapable of living independently (modified Rankin score ≥3).
9. The survival expectation is less than 1 year.
10. All subjects who are participating in other drug/medical device clinical trials and have not completed the programme requirements
11. Inapplicable for this study at the investigators' viewpoints.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Complete aneurysm occlusion without significant parent artery stenosis (≤50%) or retreatment at 1 year post procedure | 1 year post procedure
  Proportion of subjects with complete occlusion of the target aneurysm, ≤50% stenosis of the parent artery at the target cerebral aneurysms at 1 year as assessed by angiography, and in whom an unplanned alternative treatment of the target cerebral aneurysms had not been performed within 1 year.
Major stroke in the territory supplied by the treated artery or neurological death at 1 year post procedure | 1 year post procedure
  National Institute of Health Stroke Scale (NIHSS) was used to assess patients after stroke in an 11-item scale with potential scores ranging from 0 to 42. Higher values represent a worse outcome. A major stroke is defined as a new neurological event which is ipsilateral and in the vascular distribution territory of the stenting procedure and that results in an increase of ≥ 4 on the NIHSS as compared to baseline.

SECONDARY OUTCOMES:
Immediate procedural success rate | Intra-procedure
  Intraoperative cerebrovascular imaging is performed to determine whether the investigational device positions exactly and covers the aneurysm neck effectively.
Complete aneurysm occlusion rate at 180 days and 1 year post procedure | 180 days, 1 year post procedure
  Complete occlusion was defined as complete obliteration of the aneurysm sac, including the neck (Raymond I).
Success aneurysm occlusion at 180 days and 1 year post procedure | 180 days and 1 year post procedure
  The Raymond-Roy occlusion classification (RROC) is an angiographic classification scheme for grading the occlusion of flow diverter treated cerebral aneurysms (class I: complete obliteration, class II: residual neck, class III: residual aneurysm). Higher class represent a worse outcome. The percentage of Success aneurysm occlusion in which class 1 or 2 is achieved on the Raymond Scale at the 180 days and 1 year follow-up angiographic assessments will be evaluated.
Complete aneurysm occlusion without significant parent artery stenosis (≤50%) or retreatment at 180 days post procedure | 180 days post procedure
  Proportion of subjects with complete occlusion of the target aneurysm, ≤50% stenosis of the parent artery at the target cerebral aneurysms at 180 days as assessed by angiography, and in whom an unplanned alternative treatment of the target cerebral aneurysms had not been performed within 180 days.
All-cause mortality at 30 days, 180 days and 1 year post procedure | 30 days, 180 days and 1 year post procedure
  Deaths due to any cause are calculated.
Any stroke at 30 days, 180 days and 1 year post procedure | 30 days, 180 days and 1 year post procedure
  Incidence of any stroke including ischemic and hemorrhagic stroke.
Major stroke in the territory supplied by the treated artery or neurological death at 180 days post procedure | 180 days post procedure
  National Institute of Health Stroke Scale (NIHSS) was used to assess patients after stroke in an 11-item scale with potential scores ranging from 0 to 42. Higher values represent a worse outcome. A major stroke is defined as a new neurological event which is ipsilateral and in the vascular distribution territory of the stenting procedure and that results in an increase of ≥ 4 on the NIHSS as compared to baseline.
Target aneurysmal hemorrhage at 180 days and 1 year post procedure | 180 days and 1 year post procedure
  Percentage (%) of participants who experienced a Target aneurysmal hemorrhage.
Ischemic cerebrovascular events caused by thromboembolism at 180 days and 1 year post procedure | 180 days and 1 year post procedure
  Percentage (%) of participants who experienced ischemic cerebrovascular events caused by thromboembolism.
Incidence of operation or device-related adverse events/serious adverse events during hospitalization, 30 days, 180 days and 1 year post procedure | hospitalization, 30 days, 180 days and 1 year post procedure
  Percentage (%) of participants who experienced adverse events/serious adverse events.
Rate of Device defect | within 1 year of whole trial
  Device defects refer to the unreasonable risks that may endanger human health and life safety during the normal use of medical devices in the course of clinical trials, such as label errors, quality problems, failures, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Zhang, Ph.D, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, China